CLINICAL TRIAL: NCT03738072
Title: A Study of the Effect of Intracerebral Electrical Stimulation on the Optimisation of Presurgical Planning in Drug-refractory Partial Epilepsy (StiMiC)
Brief Title: Intracerebral Electrical Stimulation and the Optimisation of Presurgical Planning in Drug-refractory Partial Epilepsy
Acronym: StiMiC
Status: Recruiting | Phase: Not Applicable | Type: Interventional
Sponsor: University Hospital, Toulouse (Other)
Responsible Party: Sponsor
Allocation: Not Applicable | Model: Single Group | Masking: None | Purpose: Diagnostic
Other Study IDs: RC31/17/0345
Record Dates: First submitted 2018-11-08; First posted 2018-11-13 (Actual); Last update posted 2024-05-08 (Actual); Status verified 2024-05

CONDITIONS: Epilepsy
Keywords: Epilepsy; Electrical Brain stimulation; Neurosurgery; stereo-electro-encephalography (SEEG)
MeSH Terms: conditions — Epilepsy

STUDY DESIGN:
Oversight: Data Monitoring Committee: No | FDA-regulated Drug: No | FDA-regulated Device: No

ARMS (1):
- StiMic stimulation condition (Experimental): StiMic stimulation condition will be evaluate during stereo-electro-encephalography and this condition will be compare to standard stimulation condition
  Interventions: Diagnostic Test: StiMiC stimulation condition

INTERVENTIONS:
Diagnostic Test: StiMiC stimulation condition — This new condition of stimulation of electrical Brain Stimulation will be evaluate to determine if this stimulation is more efficient that standard stimulation condition

SUMMARY:
Patients with drug-refractory epilepsy sometimes need to be implanted with intracerebral electrodes in order to identify their seizure onset zone. During this procedure, direct electrical brain stimulations represent a standard clinical practice to assess seizure sensitivity and for functional mapping. This study aims at assessing if extending the range of stimulation frequencies of the usual clinical frequencies is of benefit for the definition of the seizure onset zone and hence for the presurgical planning.

DETAILED DESCRIPTION:
Patients with drug-refractory epilepsy sometimes need to be implanted with intracerebral electrodes in order to identify their seizure onset zone. During this procedure, direct brain electrical stimulations is a standard clinical practice to assess seizure sensitivity and for functional mapping. However the efficiency of these stimulations can be questioned and could potentially be improved. Indeed, only two typical frequencies are commonly used in our epilepsy centre, 1Hz and 50Hz, without clear clinical or scientific justification for these specific frequencies.

This study aims at assessing if extending the range of stimulation frequencies of the usual clinical frequencies could improve the definition of the seizure onset zone and hence the presurgical planning. We will maintain the usual stimulation frequencies (standard clinical stimulations condition) and add new frequencies to the protocol (research stimulations condition). The choice of these new frequencies will be based either on the spontaneous frequency of the onset of the patients' typical seizures or on physiological frequencies depending on the brain structures stimulated (i.e., theta in the medial temporal lobe).

The protocol will be proposed to all patients undergoing a stereo-electro-encephalography (SEEG) in our epilepsy center and the efficiency of the two conditions (standard clinical stimulations condition vs research stimulations condition) will be compared. The efficiency will be assessed as any epileptic event, recorded in the intracerebral EEG or symptom induced by the stimulations. This project will last 36 months. 20 patients will be included.

ELIGIBILITY:
Inclusion Criteria:

* all patients undergoing a stereo-electro-encephalography (SEEG), age 12 to 65 years old.

Exclusion Criteria:

* usual excluding criteria for a SEEG.

Ages: 12 Years to 65 Years | Sex: All | Healthy Volunteers: No
Age Groups: Child, Adult, Older Adult
Enrollment: 20 (Estimated)
Dates: Start 2018-11-14 (Actual); Primary Completion 2024-12 (Estimated); Study Completion 2024-12 (Estimated)

PRIMARY OUTCOMES:
Comparison of the index of efficient stimulation between standard clinical stimulation condition and StiMic stimulation condition | 22 days after implantation of electrode
  Comparison for each patient of the index of efficient stimulations (assessed as any stimulation having yielded an electrical or clinical effect over the total number of stimulations) for each condition (standard clinical stimulations condition vs research stimulations condition).

SECONDARY OUTCOMES:
efficient stimulation for each frequency of stimulation | 22 days after implantation of electrode
  Distribution of efficient stimulations (assessed as any stimulation having yielded an electrical or clinical effect) for each frequency of stimulation.
efficient stimulation for each type of brain area stimulated | 22 days after implantation of electrode
  Distribution of efficient stimulations (assessed as any stimulation having yielded an electrical or clinical effect) for each type of brain area stimulated (i.e, anatomical brain area, seizure onset zone, primary seizure propagation zone, healthy brain area or lesion).
percentage change in the neuronal discharge rate | 30 second after stimulation
  Percentage change in the neuronal discharge rate 30 seconds after the stimulation compared to the 30 seconds before the stimulation, depending on the frequency of stimulations.
percentage change in the neuronal discharge rate for stimic stimulation condition | 30 second after stimulation
  Percentage change in the neuronal discharge rate 30 seconds after the stimulation compared to the 30 seconds before the stimulation, depending on the effect of the stimulation (electrical or clinical as defined in the primary outcome)

CONTACTS AND LOCATIONS:
Overall Officials: Jonathan Curot, MD, Principal Investigator — CHU of Toulouse
Locations (1):
- CHU de Toulouse, Toulouse, France

IPD SHARING:
Plan to Share IPD: No